CLINICAL TRIAL: NCT00587002
Title: Differences in Epicardial Plaque and Microvascular Function in Women With an Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Patricia Best, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-001023; Epi-Plaque
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Myocardial Infarction
Keywords: Acute Coronary Syndrome; Women
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Gender comparison
  Interventions: Procedure: IVUS

INTERVENTIONS:
Procedure: IVUS — Intravascular ultrasound with virtual histology

SUMMARY:
The broad objective is to advance our understanding of both in vivo anatomical and functional changes that are present in the coronary arteries in women who have an acute coronary syndrome. Specific focus will be placed on the age of the women as there may be distinct differences in younger women (< 50 years) given the marked increase in mortality in this population.

DETAILED DESCRIPTION:
The hypothesis of the current study is that plaque erosion and microvascular dysfunction are key features responsible for the increased peri-MI mortality in young women. In order to test this hypothesis the following specific aims are proposed using a special intravascular ultrasound technique called virtual histology and microvascular function (effect of intracoronary adenosine on coronary blood flow) in patients coming to the cardiac catheterization laboratory with an acute MI:

1. To determine if plaque rupture or plaque erosion is more prevalent in young women (<50 years) compared with older women (≥ 50 years) and men in the development of an acute MI
2. To determine if inflammatory mediators of plaque rupture are higher in older women and men with an acute MI compared with younger women
3. To determine if microvascular function is abnormal in young women undergoing percutaneous coronary revascularization with an acute MI compared to older women and men
4. To determine if alterations exist in the number and function of EPCs in young women (<50 years) compared with older women (≥ 50 years) and men who have had an acute MI and to determine the association with microvascular function

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Acute coronary syndrome defined as at least two of the following:

A) an elevated cardiac biomarker (troponin or CK-MB), B) new or dynamic ECG changes in at least 2 contiguous standard electrocardiographic leads of ST depression > 1 mm or ST elevation of >1 mm or T-wave inversions, C) chest pain or discomfort of at least 15 minutes duration, D) a new wall motion abnormality by echocardiography

* Patient who is undergoing coronary angiography
* Physician planning to perform IVUS for treatment of the infarct-related vessel

Exclusion Criteria:

* Creatinine > 2.0 mg/dL (most recent)
* Hemodynamically unstable patients (systolic blood pressure < 90 mmHg or heart rate > 110 beats/ minute or presence of an intra-aortic balloon pump)
* Coronary revascularization (percutaneously or surgically) within 6 months
* The use of chronic immunosuppressive agents
* No target lesion was found at the time of cardiac catheterization that will be percutaneously intervened upon (the patient must undergo percutaneous coronary intervention)
* Inability to give informed consent
* Pregnant or lactating women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Plaque Virtual Histology | Performed during PCI

SECONDARY OUTCOMES:
Endothelial Progenitor Cells | Collected immediately pre PCI
Microvascular function in the noninfarct related vessel | Assessed immediately post PCI
Virtual Histology in noninfarct related vessel | Assessed immediately post PCI

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Best, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States